CLINICAL TRIAL: NCT02832791
Title: Comparative Study of Anterior Cruciate Ligament Reconstruction Using Quadriceps Tendon Versus Hamstring Tendon in Postoperative Clinical and Functional State: a Prospective Randomized Controlled Study
Brief Title: Comparative Study of Anterior Cruciate Ligament Reconstruction (Quadriceps Versus Hamstring Tendon)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P16-R13
Record Dates: First submitted 2016-07-06; First posted 2016-07-14 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Acute Injury of Anterior Cruciate Ligament
Keywords: ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION; QUADRICEPS TENDON; HAMSTRING TENDON

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QUADRICEPS TENDON (Active Comparator): ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION USING QUADRICEPS TENDON
  Interventions: Procedure: QUADRICEPS TENDON
- HAMSTRING TENDON (Active Comparator): ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION USING HAMSTRING TENDON
  Interventions: Procedure: HAMSTRING TENDON

INTERVENTIONS:
Procedure: QUADRICEPS TENDON — Once the limb is prepped and draped,it is exsanguinated, and the tourniquet is raised to 250 mm Hg. We will make an arthroscopic examination through an anterolateral viewing portal to corroborate the ACL injury as well as the determination of possible associated lesions. The accessory medial portal is stablished slightly above the joint line (about 2 cm of the medial edge of the patel) that is used as an instrumentation portal. Then,, a high anteromedial portal, is made higher than the previous to see the femoral footprint. Once the associated meniscal or cartilaginous lesions are addressed attention turns to the harvesting of the graft. A 4 cm vertical incision is made starting at the proximal pole of the patella and directed proximally and centered in line with the quadriceps tendon. The subcutaneous tissue is dissected and a 70-80 mm long ,10 mm wide and 7mm depth graft is obtained with the use of a n21 scalpel 2cm of both limbs of the graft are sutured
  Other Names: quadriceps tendon graft
  Arms: QUADRICEPS TENDON
Procedure: HAMSTRING TENDON — Once the limb is prepped and draped,it is exsanguinated, and the tourniquet is raised to 250 mm Hg. The procedure begins with an arthroscopic examination through an anterolateral viewing portal to corroborate the ACL injury as well as the determination of possible associated lesions. The accessory medial portal is stablished slightly above the joint line, at about 2 cm of the medial edge of the patellar tendon. This portal is used as an instrumentation portal. A third portal, a high anteromedial portal, is made higher than the previous, this portal will allow visualization of the femoral footprint.
  Once the associated meniscal or cartilaginous lesions are addressed attention turns to the harvesting of the graft.
  A 4cm oblique incision is made starting 2 cm medial to the tibial tubercle and directed proximally and medially. After dissecting the subcutaneous tissue the Sartorius fascia is incised and both tendons are identified and harvested with the use of a tendon stripper
  Other Names: hamstring tendon graft
  Arms: HAMSTRING TENDON

SUMMARY:
The purpose of this randomized study is to compare clinical and functional outcomes of both surgery techniques for anterior cruciate ligament reconstruction (using quadriceps tendon versus hamstring tendon) after reconstruction in athletes.

DETAILED DESCRIPTION:
Background: The anterior cruciate ligament (ACL) is the most commonly injured ligament of the knee. An ACL-deficient knee can lead to recurrent instability, meniscus tears, and osteoarthritis. Patients treated with an ACL reconstruction (ACLR) have long term success rates of 80 percent to 95 percent. Graft selection may influence outcomes following ACLR. Despite the popularity of the procedure, the preferred graft remains controversial. In the past, bone-patellar tendon-bone grafts have been considered the gold-standard surgical option. However, concerns regarding donor-site morbidity have led to a shift in practice by many surgeons to use quadruple hamstring tendons (HT).Several studies have shown a deficit in the quadriceps and the hamstrings strength after using HT as a graft for ACLR . Recently, there has been an increased interest in the quadriceps tendon as graft option for ACL reconstruction. The benefits of quadriceps tendon autograph include advantageous biomechanical properties, preservation of hamstring anatomy and function, as well as a reduced incidence of donor-site morbidity. To our knowledge there is no randomized controlled trial in the literature comparing QT and HTas autografts for ACLR.

Objective: The purpose of this randomized prospective study is to compare clinical and functional outcomes after using the QT and HT tendons for ACL reconstruction in athletes.

Methods: 55 athletes patients will be recruited from Martín Gómez Clinic from Granada (Spain) and Nutuality of footballers from Andalusian (Spain). Patients will be randomized in two groups: quadriceps tendon versus hamstring tendon. Clinical and functional outcomes will be measured before surgery and three and six months after that. All patients will be operated on by the same senior surgeon and both group will received the same postoperative rehabilitation protocol. Prior to the surgery the participants or their legal representatives must sign the informed consent for participation in this research.

Discussion: The benefits of ACL reconstruction surgery show enough scientific evidence that justifying the emergence of new procedures that improve the outcome of the surgery and the reduction of possible comorbidities. The high prevalence of this disease and the therapeutic success of ACL reconstruction makes that there is an increase of the number of subjects who have received this treatment. However, there is not enough randomized trials that examines the different techniques in terms of clinical and functional outcomes or the risk of comorbidities.

Subjects were placed in the upright position with the hip flexed at 90°. To determine the height of the chair, the lateral femoral condyle was aligned with the rotational axis of the dynamometer. Before each test, the patient was instructed to perform 3 practice repetitions. The highest peak torque value for each velocity was determined, compared to the uninjured side, and described as percent of knee extensor and flexor muscles strength deficits.

ELIGIBILITY:
Inclusion Criteria:

* Ages: < 40 years old
* Genders eligible for Study: both

Exclusion Criteria:

* LCA injury diagnosis base on clinical and radiographic features with less than 6 months of evolution of the lesion at diagnosis time.
* Recreational or federated athletes

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Isokinetic strenght: | Patients will be followed over 2 years
  the assessment will be made with GENU 3 dynamometer (GENU 3, Easytech, Firenze, Italy), using isokinetic parameters at angular velocities of 60°/sec (3 repetitions), 180°/sec (5 repetitions) and 300°/sec (15 repetitions) with 30 seconds of rest among these. To determine the height of the chair, the lateral femoral condyle was aligned with the rotational axis of the dynamometer. The peak torque, average torque and flexor-extensor torque rate value. Patients will be warm up in a cycle ergometer previously (5 min) and them performing mobilization exercises and stretching in lower limbs (5 min).

SECONDARY OUTCOMES:
Visual Analogical Scale (VAS) | Patients will be followed over 2 years
  the participants will be completed a visual analogue scale (0-10 points) to assess the presence of knee pain.
Pressure Pain Thresholds: | Patients will be followed over 2 years
  We will use an electronic algometer (Somedic AB, Farsta, Sweden) over 6 points: epicondyle (1), at the midpoint between the greater trochanter and the lateral condyle of the femur on the external (2), at three centimeters above the patella in the vastus medialis (3), at the midpoint between the lower pole of the patella and the anterior tuberosity of the tibia (4), at 3 cm above the patella in midline of the thigh (5) and at the inclusion of the goose leg. The mean of 3 trials will be used for the main analysis.
MUSCLE ARQUITECTURE | Patients will be followed over 2 years
  an ultrasound device (MyLab™ 25, Esaote Medical Systems,Genova, Italy) and a 12 MHz linear probe will be used in this study. The depth and width of quad tendon and articular cartilage of femoral trochlea will be captured.
ANTEROPOSTERIOR LAXITY | Patients will be followed over 2 years
  it will be measured using the KT-2000 TM arthrometer (MEDmetric, Sn Diego, CA, USA)
Tegner questionnaire | Patients will be followed over 2 years
  It is a subjective satisfaction index of on a scale of 0 to 100
Single-legged hop test | Patients will be followed over 2 years
  The patient is placed standing on one leg and must jump as far as possible landing on the same leg.

OTHER OUTCOMES:
Body Mass Index | Patients will be followed over 2 years
  in kg/m2, will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)
Fat mass | Patients will be followed over 2 years
  %fat mass will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)
Lean Mass | Patients will be followed over 2 years
  kg of lean mass will be assessed by with bioelectrical impedance analysis (Inbody 720; Biospace, Seoul, South Korea)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Martín-Alguacil, Study Chair — Martín Gómez Clinic from Granada (Spain) and Nutuality of footballers from Andalusian (Spain)
Locations (1):
- Facultad Ciencias de la Salud, Granada, Spain